CLINICAL TRIAL: NCT00669461
Title: Lubiprostone as a Treatment for Constipation in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Arkansas (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 78055; 78055; FWA00001119
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Constipation; Parkinson's Disease
Keywords: Constipation; Parkinson's Disease
MeSH Terms: conditions — Constipation; Parkinson Disease | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental)
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — Lubiprostone 24 mcg BID orally for 4 weeks

SUMMARY:
Delayed colonic transient time secondary to a multi-degenerative process is the most likely cause of constipation in idiopathic PD. Since lubiprostone demonstrated its ability to accelerate colonic transit time in healthy volunteers in addition to activating the chloride channels in the intestinal cells, it has the potential to improve constipation in patients with PD with no subsequent adverse events on the control of the neurological manifestation of PD. So we hypothesize the following:

1. Lubiprostone will improve ratings on the Bristol stool form scale (BSFS) in patients with PD induced constipation compared to baseline.(primary)
2. Lubiprostone will increase the number of spontaneous bowel movements (SBM) per week, compared to baseline. (secondary)
3. Lubiprostone will improve health related quality of life in subjects with PD induced constipation. ( secondary)

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-85 years
2. Diagnosis of Parkinson's disease
3. Constipation as defined by the Rome III committee
4. BSFS of more or equal to 1 and less or equal to 3
5. Normal colonoscopy in the last 5 years( normal defined as absence of obstructive lesions in the colon)
6. All women subjects will be post menopausal or surgically sterile.

Exclusion Criteria:

1. Known hypersensitivity reaction to Amitiza ( Lubiprostone)
2. Known significant adverse effects to previous treatment with Lubiprostone which include; new or worsening abdominal pain, severe diarrhea, nausea, vomiting, and severe headache.
3. Renal dysfunction with creatinine clearance less than 15 ml/min
4. Abnormal liver enzymes or history of chronic liver disorder
5. History of bowel obstruction, , or abdominal adhesions .
6. Abnormal Colonoscopy ( obstructive lesions within the colon)
7. Inability to give informed consent

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhannad M Heif, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lubiprostone: patient received treatment( lubiprostone)24 mcg po BID for 4 weeks
Period: Overall Study
Arm/Group | Lubiprostone
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lubiprostone
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (0)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Bristol Stool Form Scale (BSFS) at Baseline, End of 4 Weeks and End of 6 Weeks
Description: The average BSFS will be determined at baseline (prior to the start lubiprostone) and compared with average rating of BSFS at end of the 4 weeks of treatment with Lubiprostone and at end of 2 weeks after stopping the Lubiprostone. BSFS is scale between 1-7, it measured the shape of the stool. BSFS is a scale between 1-7, where 1 correlates with the firmest stool and 7 correlates with entirely liquid stool. Measure was reported at end of week #1-Baseline-,end of Week #5 ( after taking the lubiprostone for 4 weeks) and end of week # 7 ( end of 2 weeks after stopping the Lubiprostone).
Time Frame: up to 6 weeks
Population: Analysis was not performed for this outcome measure secondary to the small sample size ( one patient)
Groups:
- Lubiprostone: Lubiprostone 24 micrograms po BID given for total of 4 weeks
Arm/Group | Lubiprostone
Number analyzed (Participants) | 0

2. Secondary Outcome: Average Number of Spontaneous Bowel Movements (SBM) Per Week
Description: Average number of spontaneous bowel movements (SBM) per week,measured at baseline, at end of 4 weeks of treatment with Lubiprostone and at 2 weeks after stopping Lubiprostone (( so measure was reported at end of week # 1-Baseline-,end of Week #5 ( after taking the lubiprostone for 4 weeks) and end of week # 7 ( end of 2 weeks after stopping the Lubiprostone)).
Time Frame: up to 6 weeks
Population: Analysis was not performed for this outcome measure secondary to the small sample size ( one patient.
Arm/Group | Lubiprostone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Arm/Group | Lubiprostone
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes